CLINICAL TRIAL: NCT05733312
Title: Intraoperative Evaluation of Focused Ultrasound-induced Blood-brain Barrier Disruption
Brief Title: Extracellular Impact of Ultrasound-induced Blood-brain Barrier Disruption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-001933; NCI-2024-03111 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-01-28; First posted 2023-02-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Focused Ultrasound (Experimental): Subjects with known or suspected glioma (≥3cm) undergoing routine planned neurosurgical resection will undergo a focused ultrasound prior to the surgery with the InSightec's ExAblate Neuro Model 4000 Type 2.0 (220 KHz) system
  Interventions: Device: InSightec's ExAblate Neuro Model 4000 Type 2.0 (220 KHz) system

INTERVENTIONS:
Device: InSightec's ExAblate Neuro Model 4000 Type 2.0 (220 KHz) system — Focused ultrasound which targets energy to a specific area in the brain based on imaging and disrupts the blood brain barrier which keeps certain drugs and other molecules out of the brain.

SUMMARY:
This study seeks to determine the impact of focused ultrasound (FUS) on the composition of the tumor extracellular microenvironment. Researchers will evaluate regions that are very abnormal, as well as regions that have less evidence of disease. A sub-portion of each of these areas will be targeted by focused ultrasound. Microdialysis catheters will then be placd into each region that has and has not been exposed to FUS (total of 4 catheters) to determine how FUS impacts the the brain and tumor extracellular metabolome, including concentration of routine drugs systemically administered prior to, and during surgery. Researchers hope that this information will help reveal the relative contribution of blood-derived compounds to the tumor microenvironment. If successful, microdialysis could be leveraged in the future to simultaneously evaluate pharmacokinetic and pharmacodynamic impacts of future candidate therapies, including those delivered with the aid of FUS.

DETAILED DESCRIPTION:
This protocol performs FUS immediately prior to clinically indicated brain tumor resection. Accordingly, any drugs administered in the context of routine clinical care, such as Ancef, levetiracetam, and mannitol) and imaging agents (gadolinium and iopamidol) clinically available for pre-operative imaging via MRI or CT, respectively, will be quantified in plasma as well as the interstitial fluid of brain tumor and adjacent brain tissue within and outside the volume of FUS treatment. Patients with large (≥3cm) gliomas and no known contraindications to contrast agents or surgery will be recruited to undergo pre-operative Exablate 4000 Type-2 MR-guided FUS prior to intraoperative high molecular weight microdialysis and standard-of-care glioma resection. Intra-operative CT or O-arm will be obtained with contrast to document the location of catheters relative to tumor and region of blood brain barrier disruption following FUS prior to tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic evidence suggesting a diagnosis of a diffuse glioma, or a prior diagnosis of a diffuse glioma, which is large enough (≥3cm) for half of the tumor to be targeted by FUS, but small enough for the standard-of-care resection to incorporate some regions of relatively normal brain adjacent to tumor.
* Planned neurosurgical resection of this suspected or previously diagnosed brain tumor as part of routine clinical care.
* Provide written informed consent for the current study and the Neuro-Oncology biorepository for archiving of microdialysate and blood samples collected on this protocol.
* ECOG performance status (PS) 0, 1, or 2. Willing to undergo neurosurgical resection at Mayo Clinic (Rochester, MN).

Exclusion Criteria:

* Patients who are not appropriate surgical candidates due to current or past medical history or uncontrolled concurrent illness which limits safety of or compliance to study proceedings.
* Vulnerable populations: pregnant or nursing women, prisoners, mentally handicapped.
* Contraindication to Definity®.
* Cardiac disease or coagulative disease (such as cerebral or systemic vasculopathy, abnormal platelets, documented MI within 6 months of enrollment, pacemaker, hemodynamically unstable cardiac arrhythmia, unstable congestive heart failure, or left ventricular ejection fraction <50%), that would preclude the use of Definity ®, FUS-induced BBB disruption, or surgical resection.
* Any blood-borne infection that may lead to meningitis or brain abscess due to BBB-disruption.
* Active seizure disorder that is not attributable to the patient's tumor which is not controlled by medication or due to active drug or alcohol disorder which may be worsened by BBB-disruption.
* Patients for whom the surgeon feels 5-ALA would be required to perform an optimal resection, since 5-ALA will not be permitted for patients participating in this study.
* Patients who are at risk of FUS-related complications due to potential risks associated with skull anatomy as determined by pre-operative CT assessment, based on skull thickness, curvature, density, or other features that would increase the risk of skull complications with FUS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 3 months post-surgery
  Number of adverse deemed related to FUS and/or intraoperative microdialysis after the integration of FUS and intraoperative microdialysis into the neurosurgical workflow for tumor resection
Number of microdialysate aliquots | 3 months post-surgery
  Number of microdialysate aliquots collected containing >10 μL of volume

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials